CLINICAL TRIAL: NCT06722963
Title: Comparison of the Efficacy of Intraperitoneal Instillation of Fentanyl Versus Nalbuphine As Adjuvants to Bupivacaine for Postoperative Pain Relief in Patients Undergoing Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sameh Saad Reyad, Resident Doctor at Anesthesia and Intensive Care Department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: fentanyl vs nalbuphine cholecy
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: fentanyl; nalbuphine
MeSH Terms: interventions — Fentanyl; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent anesthesiologist randomly divided the patients into 35 groups of patients each using computer-generated random numbers fentanyl group and nalbuphine group (Group F and Group N). We discreetly placed the randomization results in envelopes until the end of the study. Both nalbuphine and fentanyl are colorless liquids, and they were digitally encoded so that the researchers who were responsible for postoperative follow-up and data processing were blinded to the group allocation during the whole study period. All patients were also blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fentanyl group (Experimental): Fentanyl used as an adjuvant to bupivacaine for intraperitoneal instillation during laparoscopic cholecystectomy, a dose is 50 micrograms is commonly added to the local anesthetic solution.
  Interventions: Drug: fentanyl
- Nalbuphine group (Experimental): patients will receive Nalbuphine in a Doses ranging from 10 mg have been studied as adjuvants to bupivacaine
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: fentanyl — Fentanyl used as an adjuvant to bupivacaine for intraperitoneal instillation during laparoscopic cholecystectomy, a dose is 50 micrograms is commonly added to the local anesthetic solution.
  Arms: Fentanyl group
Drug: Nalbuphine — Nalbuphine in doses ranging from 10 mg have been studied as adjuvants to bupivacaine
  Arms: Nalbuphine group

SUMMARY:
Given the complexity of postoperative pain following laparoscopic surgery, specialists recommend a multimodal approach to effective analgesic management . The origin of pain after LC is multifactorial and complex in nature. Pain arising from incision sites is parietal pain, whereas pain from the gall bladder bed is mainly visceral in nature, and shoulder pain is mainly referred owing to the residual CO2 irritating the diaphragm. Various strategies have been employed for pain relief after laparoscopic procedures, including the use of intraperitoneal local anesthetics, either alone or in combination with opioid analgesics.

the efficacy of intraperitoneal instillation of fentanyl versus nalbuphine as adjuvants to Bupivacaine for postoperative pain relief in patients undergoing laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is recognized as the gold standard for managing gallbladder stones due to its numerous advantages over open surgery . These benefits include quicker and easier recovery, reduced operative morbidity, less postoperative pain, shorter convalescence, and overall lower costs

Intraperitoneal administration of local anesthetics is used by many surgeons as a method to provide effective pain relief while minimizing the adverse effects of systemic analgesics, including NSAIDs and opioids. The rationale for this route of administration is that the local anesthetics will block the visceral nociceptive conduction from peritoneum. In addition, systemic absorption from the large peritoneal surface may occur, providing additional mechanism of analgesia . This technique was first evaluated in patients undergoing gynecological laparoscopy and showed reduction in postoperative shoulder pain . With the possibility that a similar analgesic effect might be achieved in LC, several trials assessing the efficacy of Intraperitoneal local anesthetics in LC were carried out with conflicting results, regarding severity of postoperative pain, duration of analgesia, and total analgesic consumption in 24 h. The difference in outcome of studies on instillation of local anesthetics may result from dose, volume, or concentration of the drug; timing of instillation (before or after surgery); site of administration (subdiaphragmatic, over gall bladder bed, and/or port infiltration); and instillation in Trendelenberg's versus supine position .

Fentanyl and nalbuphine are two widely used opioids considered for pain management . Fentanyl is a potent synthetic opioid similar to morphine but produces analgesia to a greater extent. This robust pharmacologic agent is typically 50 to 100 times more potent than morphine . it is renowned for its rapid onset and strong analgesic properties. It is extensively used in clinical settings to manage acute pain .

On the other hand, nalbuphine, a mixed agonist-antagonist opioid, acts as an antagonist at μ-receptors and agonist at k-receptors that work reasonably potent analgesia. It offers effective pain relief, particularly with a lower risk of respiratory depression. It also provides prolonged analgesia and is associated with fewer side effects, such as pruritus, nausea, and vomiting, than fentanyl .

This route of administration is noninvasive, simple to perform, does not involve additional neuraxial block, and is particularly suited for the practice of ambulatory anesthesia. However, duration of analgesia may be limited for few hours. So, addition of adjuvants such as narcotics, α2 agonists, or NSAIDs has been proposed to prolong the postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Both sex
* Patients who were in risk-scoring groups I-II of the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* • Patient's refusal.

  * body mass index (BMI) ≥40 kg/m2.
  * History of hypersensitivity to the drugs being evaluated
  * Inability to comprehend postoperatively the pain assessment scale/neuropsychiatric disorders.
  * chronic use of opioids and opioid addiction
  * Patients with acute cholecystitis
  * Carcinoma of gall bladder
  * Pregnant female
  * Bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
time to first analgesic request | 24 hours
  comparison of the post-operative analgesic effect regarding the time to first analgesic request of fentanyl versus nalbuphine as adjuvants to Bupivacaine in patients undergoing laparoscopic cholecystectomy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laisalmi M, Koivusalo AM, Valta P, Tikkanen I, Lindgren L. Clonidine provides opioid-sparing effect, stable hemodynamics, and renal integrity during laparoscopic cholecystectomy. Surg Endosc. 2001 Nov;15(11):1331-5. doi: 10.1007/s004640090126. Epub 2001 Aug 16. PMID 11727145
- [Background] Khodorova A, Navarro B, Jouaville LS, Murphy JE, Rice FL, Mazurkiewicz JE, Long-Woodward D, Stoffel M, Strichartz GR, Yukhananov R, Davar G. Endothelin-B receptor activation triggers an endogenous analgesic cascade at sites of peripheral injury. Nat Med. 2003 Aug;9(8):1055-61. doi: 10.1038/nm885. Epub 2003 Jun 29. PMID 12847519
- [Background] Kuhry E, Jeekel J, Bonjer HJ. Effect of laparoscopy on the immune system. Semin Laparosc Surg. 2004 Mar;11(1):37-44. doi: 10.1177/107155170401100107. PMID 15094977